CLINICAL TRIAL: NCT07261826
Title: Real-World Study on Fecal Microbiota Transplantation: Long-Term Effectiveness and Safety Statistics
Status: Recruiting | Type: Observational
Sponsor: Chen QiYi (Other)
Responsible Party: Sponsor-Investigator, Chen QiYi, Chief of Functional Gastrointestinal Surgery, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: SHSY-IEC-6.0/25K221/P01
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Clostridium Difficile Infection Recurrence; Ulcerative Colitis (UC); Crohn Disease (CD); Irritable Bowel Syndrome (IBS); Chronic Functional Constipation; Chemotherapy-Induced Colitis; PD-1 Associated Enteritis; Autism Spectrum Disorder; Incomplete Intestinal Obstruction
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Irritable Bowel Syndrome; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (9):
- Clostridium Difficile Infection Recurrence
- Ulcerative Colitis (UC)
- Crohn Disease (CD)
- Irritable Bowel Syndrome (IBS)
- chronic functional constipation
- Chemotherapy-Induced Colitis
- PD-1 associated enteritis
- Autism Spectrum Disorder
- incomplete intestinal obstruction

SUMMARY:
This is a large-scale observational study aiming to evaluate the long-term effectiveness and safety of Fecal Microbiota Transplantation (FMT). FMT is a procedure that transfers gut bacteria from healthy donors to patients to restore a balanced gut microbiome.

The study will follow approximately 4,000 patients who have received or will receive FMT for conditions like recurrent C. difficile infection, inflammatory bowel disease, functional gastrointestinal disorders, and certain neurological conditions.

The main goals are to:

* Assess the disease remission rates at 3 months, 1 year, and 5 years after FMT.
* Monitor the long-term safety and any potential side effects.
* Identify factors that may influence how well a patient responds to the treatment.

This research will use both existing patient data (retrospective cohort) and newly collected data from future patients (prospective cohort). The findings are expected to help improve and standardize FMT treatment for better patient care.

DETAILED DESCRIPTION:
This is a single-center, real-world observational study combining retrospective and prospective cohorts to systematically evaluate the long-term effectiveness and safety of Fecal Microbiota Transplantation (FMT).

The study plans to enroll approximately 4,000 patients who have undergone FMT for a range of diseases, including recurrent Clostridium difficile infection, inflammatory bowel disease, functional gastrointestinal diseases, and certain extra-intestinal disorders.

The primary objective is to assess the real-world clinical remission rates at 3 months, 1 year, and 5 years post-FMT. Secondary objectives include evaluating long-term safety and adverse events, measuring improvements in quality of life, and exploring factors (such as delivery route, donor selection, and patient characteristics) that predict treatment success. Data will be collected from medical records and through planned follow-up visits. Advanced statistical and machine learning models will be used to analyze the data and build predictive models.

The results of this large-scale study will provide high-quality evidence to support the standardized and precise clinical application of FMT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with one of the target diseases.
* Age ≥ 3 years.
* Have received at least one Fecal Microbiota Transplantation (FMT) treatment.
* Availability of complete baseline and follow-up data for analysis.
* Provide signed informed consent (for the prospective cohort) OR consent for the use of clinical data (for the retrospective cohort).

Exclusion Criteria:

* Clinical data is severely missing, making efficacy assessment impossible.
* Presence of severe complications that may jeopardize safety or confound the study results.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of approximately 4,000 patients who have undergone Fecal Microbiota Transplantation (FMT) at our center. This includes a retrospective cohort of about 3,000 patients treated between January 2017 and August 2025, whose data will be collected from medical records, and a prospective cohort of about 1,000 new patients to be enrolled from September 2025 to June 2028.
  Participants must be ≥3 years of age and diagnosed with one of the target diseases, including but not limited to recurrent Clostridium difficile infection, inflammatory bowel disease, functional gastrointestinal disorders, and certain extra-intestinal diseases. All participants must have received at least one FMT treatment and have available baseline data.
  This real-world study aims to include a broad patient population reflective of routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
8-Week Clinical Cure of Recurrent CDI | 8 weeks after the final FMT treatment
  Percentage of participants with sustained clinical cure at 8 weeks post-treatment, defined as persistent resolution of diarrhea (formed stools <3 times per day) AND a negative test for C. difficile toxin.
Treatment Response in Chronic Constipation at 8 Weeks | 8 weeks after the final FMT treatment
  Percentage of participants meeting all of the following criteria at 8 weeks: >3 complete spontaneous bowel movements per week, Bristol Stool Form Scale (BSFS) type 3-5, and a reduction of >30% in the Patient Assessment of Constipation Symptoms (PAC-SYM) score.
Corticosteroid-Free Clinical Remission in IBD at 8 Weeks | 8 weeks after the final FMT treatment
  Percentage of participants achieving corticosteroid-free clinical remission. For Ulcerative Colitis (UC), defined as a Mayo score ≤2 with no subscore >1. For Crohn's Disease (CD), defined as a Crohn's Disease Activity Index (CDAI) score <150.
Symptom Relief in IBS at 3 Months | 3 months after the final FMT treatment
  Percentage of participants experiencing relief of abdominal pain or discomfort related to defecation for 3 consecutive months, with stool consistency rated as Bristol Stool Form Scale (BSFS) type 3-5.
Treatment Response in Autism at 12 Weeks | 12 weeks after the final FMT treatment
  Percentage of participants meeting the response criteria at Week 12, defined as an Autism Behavior Checklist (ABC) score <31 AND a score of 1 (very much improved) on the Clinical Global Impression-Improvement (CGI-I) scale.
Symptom Improvement in Incomplete Bowel Obstruction | 8 weeks after the final FMT treatment
  Percentage of participants achieving a reduction of >50% in abdominal distension and/or pain, AND weaning off parenteral nutrition.
Symptom Resolution in Drug-Induced Enteritis | 8 weeks after the final FMT treatment
  Percentage of participants achieving symptom resolution, defined as a reduction to CTCAE grade ≤1 (stool frequency increase <4 times per day from baseline, without abdominal pain, hematochezia, or mucus), AND requiring corticosteroids <10 mg prednisone equivalent per day.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Rupnik M, Wilcox MH, Gerding DN. Clostridium difficile infection: new developments in epidemiology and pathogenesis. Nat Rev Microbiol. 2009 Jul;7(7):526-36. doi: 10.1038/nrmicro2164. PMID 19528959
- [Result] Khoruts A, Sadowsky MJ. Understanding the mechanisms of faecal microbiota transplantation. Nat Rev Gastroenterol Hepatol. 2016 Sep;13(9):508-16. doi: 10.1038/nrgastro.2016.98. Epub 2016 Jun 22. PMID 27329806
- [Result] EISEMAN B, SILEN W, BASCOM GS, KAUVAR AJ. Fecal enema as an adjunct in the treatment of pseudomembranous enterocolitis. Surgery. 1958 Nov;44(5):854-9. No abstract available. PMID 13592638
- [Result] Zhang F, Luo W, Shi Y, Fan Z, Ji G. Should we standardize the 1,700-year-old fecal microbiota transplantation? Am J Gastroenterol. 2012 Nov;107(11):1755; author reply p.1755-6. doi: 10.1038/ajg.2012.251. No abstract available. PMID 23160295
- [Result] Petersen C, Round JL. Defining dysbiosis and its influence on host immunity and disease. Cell Microbiol. 2014 Jul;16(7):1024-33. doi: 10.1111/cmi.12308. Epub 2014 Jun 2. PMID 24798552
- [Result] Baumler AJ, Sperandio V. Interactions between the microbiota and pathogenic bacteria in the gut. Nature. 2016 Jul 7;535(7610):85-93. doi: 10.1038/nature18849. PMID 27383983
- [Result] Zheng D, Liwinski T, Elinav E. Interaction between microbiota and immunity in health and disease. Cell Res. 2020 Jun;30(6):492-506. doi: 10.1038/s41422-020-0332-7. Epub 2020 May 20. PMID 32433595
- [Result] Rowland I, Gibson G, Heinken A, Scott K, Swann J, Thiele I, Tuohy K. Gut microbiota functions: metabolism of nutrients and other food components. Eur J Nutr. 2018 Feb;57(1):1-24. doi: 10.1007/s00394-017-1445-8. Epub 2017 Apr 9. PMID 28393285
- [Result] Qin J, Li R, Raes J, Arumugam M, Burgdorf KS, Manichanh C, Nielsen T, Pons N, Levenez F, Yamada T, Mende DR, Li J, Xu J, Li S, Li D, Cao J, Wang B, Liang H, Zheng H, Xie Y, Tap J, Lepage P, Bertalan M, Batto JM, Hansen T, Le Paslier D, Linneberg A, Nielsen HB, Pelletier E, Renault P, Sicheritz-Ponten T, Turner K, Zhu H, Yu C, Li S, Jian M, Zhou Y, Li Y, Zhang X, Li S, Qin N, Yang H, Wang J, Brunak S, Dore J, Guarner F, Kristiansen K, Pedersen O, Parkhill J, Weissenbach J; MetaHIT Consortium; Bork P, Ehrlich SD, Wang J. A human gut microbial gene catalogue established by metagenomic sequencing. Nature. 2010 Mar 4;464(7285):59-65. doi: 10.1038/nature08821. PMID 20203603